CLINICAL TRIAL: NCT00441454
Title: Retropubic vs. Transobturator Tension-free Vaginal Tape (TVT vs. TVT-O): A Randomized Trial
Brief Title: Retropubic vs. Transobturator Tension-free Vaginal Tape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Urogynecology Working Group (AUWG) (Other)
Responsible Party: Principal Investigator, Karl Tamussino, MD, PI, Austrian Urogynecology Working Group (AUWG)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVT vs. TVT-O
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; surgery; tension-free vaginal tape; retropubic; transobturator; quality-of-life
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (2):
- A (Active Comparator): Retropubic Tension-free Vaginal Tape (TVT)
  Interventions: Device: Retropubic Tension-free vaginal tape (TVT)
- B (Active Comparator): Transobturator Tension-free Vaginal Tape (TVT-O)
  Interventions: Device: Transobturator Tension-free vaginal tape (TVT-O)

INTERVENTIONS:
Device: Transobturator Tension-free vaginal tape (TVT-O) — tension-free vaginal tape (TVT)
  Arms: B
Device: Retropubic Tension-free vaginal tape (TVT) — Retropubic Tension-free vaginal tape (TVT)
  Arms: A

SUMMARY:
The so-called tension-free vaginal tape (TVT), first described in Sweden in 1996, has become a standard operation worldwide for the treatment of women with stress urinary incontinence. This tape is placed from the vagina behind the pubic bone and exits through the skin of the lower abdomen, just above the pubic bone. In 2001 a urologist in France proposed passing a similar tape laterally (as opposed to behind the pubic bone). This tape is passed through a window of the pelvic bones (the so-called obturator foramen), by what is called a transobturator approach. It is passed through the skin of the thigh (as opposed to the lower abdomen). The reason for this modification was to avoid injuring the bladder and, possibly, provide a more physiologic restoration of the continence mechanism. However, it is unclear whether the lateral (so-called transobturator approach) is as good as or better than the initial approach behind the pubic bone.

The purpose of the present study is to compare the standard (retropubic) and the newer (transobturator) approach for the placement of a tape for treating women with stress urinary incontinence.

DETAILED DESCRIPTION:
After informed consent women scheduled for surgery for stress urinary incontinence are randomized to receive a tension-free vaginal tape either by the retropubic or the transobturator approach.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery for primary stress incontinence (positive stress test at bladder filling of 300 ml) without concomitant prolapse surgery or hysterectomy
* Patient able and willing to participate in follow-up
* Informed consent

Exclusion Criteria:´

* Detrusor overactivity, predominant complaint overactive bladder (OAB)
* Major concomitant surgery
* Prolapse beyond introitus or any prolapse necessitating surgery
* Previous incontinence surgery other than colporrhaphy
* Residual urine >100 ml
* Neurologic disease
* Allergy to local anesthetic agents
* Coagulation disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2004-09; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Continence | 5 years

SECONDARY OUTCOMES:
Quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Karl F Tamussino, MD, Principal Investigator — Medical University of Graz, Dept. OB/GYN
Locations (4):
- Austria (4):
  - Dept. of Gynecology, Krankenhaus der Barmherzigen Brüder, Graz
  - Department of OB/GYN, Medical University of Graz, Graz
  - Dept. OB/GYN, Medical University of Vienna, Vienna
  - Dept. OB/GYN, Wilhelminenspital, Vienna

REFERENCES:
- [Background] de Leval J. Novel surgical technique for the treatment of female stress urinary incontinence: transobturator vaginal tape inside-out. Eur Urol. 2003 Dec;44(6):724-30. doi: 10.1016/j.eururo.2003.09.003. PMID 14644127
- [Background] Delorme E. [Transobturator urethral suspension: mini-invasive procedure in the treatment of stress urinary incontinence in women]. Prog Urol. 2001 Dec;11(6):1306-13. French. PMID 11859672
- [Background] Tamussino KF, Hanzal E, Kolle D, Ralph G, Riss PA; Austrian Urogynecology Working Group. Tension-free vaginal tape operation: results of the Austrian registry. Obstet Gynecol. 2001 Nov;98(5 Pt 1):732-6. doi: 10.1016/s0029-7844(01)01565-4. PMID 11704161
- [Background] Ulmsten U, Henriksson L, Johnson P, Varhos G. An ambulatory surgical procedure under local anesthesia for treatment of female urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):81-5; discussion 85-6. doi: 10.1007/BF01902378. PMID 8798092
- [Background] Ward K, Hilton P; United Kingdom and Ireland Tension-free Vaginal Tape Trial Group. Prospective multicentre randomised trial of tension-free vaginal tape and colposuspension as primary treatment for stress incontinence. BMJ. 2002 Jul 13;325(7355):67. doi: 10.1136/bmj.325.7355.67. PMID 12114234
- [Background] Ward KL, Hilton P; UK and Ireland TVT Trial Group. A prospective multicenter randomized trial of tension-free vaginal tape and colposuspension for primary urodynamic stress incontinence: two-year follow-up. Am J Obstet Gynecol. 2004 Feb;190(2):324-31. doi: 10.1016/j.ajog.2003.07.029. PMID 14981369
- [Derived] Tammaa A, Aigmuller T, Hanzal E, Umek W, Kropshofer S, Lang PFJ, Ralph G, Riss P, Koelle D, Jundt K, Tamussino K, Bjelic-Radisic V; Austrian Urogynecology Working Group. Retropubic versus transobturator tension-free vaginal tape (TVT vs TVT-O): Five-year results of the Austrian randomized trial. Neurourol Urodyn. 2018 Jan;37(1):331-338. doi: 10.1002/nau.23298. Epub 2017 May 2. PMID 28464312
- [Derived] Aigmuller T, Tammaa A, Tamussino K, Hanzal E, Umek W, Kolle D, Kropshofer S, Bjelic-Radisic V, Haas J, Giuliani A, Lang PF, Preyer O, Peschers U, Jundt K, Ralph G, Dungl A, Riss PA; Austrian TVT vs. TVT-O Study Group. Retropubic vs. transobturator tension-free vaginal tape for female stress urinary incontinence: 3-month results of a randomized controlled trial. Int Urogynecol J. 2014 Aug;25(8):1023-30. doi: 10.1007/s00192-014-2384-z. Epub 2014 May 13. PMID 24819327